CLINICAL TRIAL: NCT03363451
Title: A Retrospective Study on Diagnosis and Treatment of End Stage Liver Disease Complicated With Infection (SESLDIR Study)
Brief Title: A Study on Diagnosis and Treatment of End Stage Liver Disease Complicated With Infection (SESLDIR Study)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Qin Ning, Director of Department of Infectious Disease, Tongji Hospital
Other Study IDs: SESLDIR study
Record Dates: First submitted 2017-11-22; First posted 2017-12-06 (Actual); Last update posted 2018-09-14 (Actual); Status verified 2017-12

CONDITIONS: End Stage Liver Disease; Infection
MeSH Terms: conditions — End Stage Liver Disease; Infections | interventions — Anti-Bacterial Agents

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Infection Group: Patients with end stage liver disease with infection
  Interventions: Drug: Antibiotics
- Non-infection Group: Patients with end stage liver disease without infection

INTERVENTIONS:
Drug: Antibiotics — This is an observation study, no specific antibiotics will be indicated during treatment
  Groups: Infection Group

SUMMARY:
The term of End Stage of Liver Disease (ESLD) was raised in 80's of 20 Century, but without a restrict definition. Infections are the cause and effect in occurrence and development of ESLD, which not only induce or exacerbate ESLD, but also are the most combined complication. Multi-resistant bacteria, multi-organ injury, selection of anti-microbes, supporting treatment, disorder of intestine microbiota, et al are dilemma in clinical practice. Appropriate and formal diagnosis and treatment of ESLD combined infection are imperious nowadays.

ELIGIBILITY:
Inclusion Criteria:

Decompensation of liver cirrhosis:

1. ALB <35 g / L; A / G <1.0
2. TBIL> 35μmol / L;
3. ALT> 1 × ULN and / or AST> 1 × ULN
4. PTA <60%
5. Ascites or hepatic encephalopathy or esophageal variceal bleeding

Acute-on-chronic liver failure:

1. Chronic liver disease based on: chronic hepatitis or decompensated cirrhosis
2. onset time: <4 weeks
3. Hepatic encephalopathy: with or without
4. Coagulation: PTA ≤ 40% or INR ≥ 1.5
5. Jaundice: TBIL ≥ 171μmol / L or daily increase ≥ 17.1μmol / L

Chronic liver failure:

1. The basis of chronic liver disease: decompensated cirrhosis
2. onset time: -
3. Hepatic encephalopathy: with or without
4. Coagulation: PTA ≤ 40% or INR ≥ 1.5 Jaundice: significantly higher

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with chronic liver disease
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-12-30 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Complete response rate to empirical antibiotic treatment | 6 months
  The percentage of patients who achieved complete recovery from combined infection after empirical antibiotic treatment

SECONDARY OUTCOMES:
Non-liver transplant survival | 6 months
  Non-liver transplant survival rate at 30 days, 60 days and 6 months after empirical antibiotic treatment
Hospitalization time | 6 months
  Days of hospitalization after empirical antibiotic treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Infectious Disease, Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided